CLINICAL TRIAL: NCT02899195
Title: Open Label, Phase II Study of Anti - Programmed Death - Ligand 1 Antibody, Durvalumab (MEDI4736), in Combination With Chemotherapy for the First-Line Treatment of Unresectable Mesothelioma
Brief Title: Phase II MEDI4736 in Combination With Chemotherapy for First-Line Treatment of Unresectable Mesothelioma
Acronym: PrE0505
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PrECOG, LLC. (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PrE0505; ESR-15-10792 (Other: AstraZeneca)
Record Dates: First submitted 2016-09-08; First posted 2016-09-14 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Mesothelioma; Pleural Mesothelioma
Keywords: Unresectable Mesothelioma; Durvalumab; Anti-Programmed Death-Ligand 1 Antibody
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Concurrent therapy with Durvalumab, Pemetrexed and Cisplatin (or Carboplatin) for up to 6 cycles followed by Maintenance Therapy with Durvalumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab (Experimental): Pemetrexed/cisplatin will be given for up to six 3-week cycles with the addition of concurrent durvalumab every 3 weeks. The first 6 patients who are enrolled and commence treatment will be monitored for safety of the combination. Use of carboplatin in place of cisplatin will be permitted for patients who are ineligible for cisplatin due to impaired renal function at screening. For patients that receive cisplatin, carboplatin may also be substituted after Cycle 1 for cisplatin related toxicity (e.g., grade 3 ototoxicity, grade 3 nausea) at the investigator's discretion. After completion of Cycle 6 of concurrent therapy, patients with stable or responding disease per modified RECIST for malignant mesothelioma will continue on single agent durvalumab every 3 weeks until progression. Maximum duration of durvalumab treatment is 12 months starting from Cycle 1 of concurrent treatment (inclusive of any treatment delays or missed treatments).
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — On Day 1 of each 21 day cycle: Durvalumab 1120 mg IV will be administered before pemetrexed and cisplatin chemotherapy over approximately 60 minutes. Approximately 30 minutes after the durvalumab infusion is complete, pemetrexed 500 mg/m² IV will be administered over 10 minutes. Cisplatin 75 mg/m² IV over 2 hours will begin approximately 30 minutes after the end of pemetrexed administration. If carboplatin is substituted for cisplatin, carboplatin Area Under the Concentration-Time Curve (AUC) 5 will be infused over 30 minutes beginning approximately 15-30 minutes after the end of the pemetrexed administration. Maintenance: On Day 1 of each 21 day cycle: Durvalumab 1120 mg IV over approximately 60 minutes.
  Other Names: MEDI4736

SUMMARY:
Patients with pleural mesothelioma that can not be surgically removed will receive durvalumab, in combination with standard chemotherapy of pemetrexed and cisplatin as first-line treatment.

Durvalumab is a type of drug called a monoclonal antibody (a type of protein). Laboratory tests show that it works by allowing the immune system to detect your cancer and reactivates the immune response. This may help to slow down the growth of cancer or may cause cancer cells to die.

The purpose of this study is to see whether adding durvalumab to standard chemotherapy will improve overall survival (OS).

DETAILED DESCRIPTION:
Mesothelioma is a malignant tumor of the mesothelial surfaces primarily arising in the thoracic pleura and is estimated to cause 43,000 deaths worldwide each year with over 3300 cases occurring annually in the United States. Approximately 80% of cases of mesothelioma are due to inflammation induced by prior asbestos exposure with a lead time from exposure to development of cancer of 20-30 years.

This is a single arm, open label phase II study of the anti-PD-L1 antibody, durvalumab, in combination with standard chemotherapy. Pemetrexed and cisplatin will be given for up to six 3-week cycles with the addition of concurrent durvalumab dosed every 3 weeks. The first 6 patients who are enrolled and commence treatment will be monitored for safety of the combination. Use of carboplatin in place of cisplatin will be permitted for patients who are ineligible for cisplatin due to impaired renal function at screening, however these patients must otherwise fulfill the eligibility criteria for the study. For patients that receive cisplatin, carboplatin may also be substituted after Cycle 1 for cisplatin related toxicity (e.g., grade 3 ototoxicity, grade 3 nausea) at the investigator's discretion. After completion of Cycle 6 of concurrent therapy, patients with stable or responding disease per modified RECIST for malignant mesothelioma will continue on single agent durvalumab every 3 weeks until progression. Maximum duration of durvalumab treatment is 12 months starting from Cycle 1 of concurrent treatment (inclusive of any treatment delays or missed treatments).

Tumor assessments will be performed approximately every 6 weeks during concurrent therapy and every 9 weeks during the maintenance phase.

Mandatory pre-treatment tumor tissue sample (i.e., obtained during a previous procedure or biopsy) and blood samples (prior to Cycle 1, Cycle 2 and Cycle 5) for research will also be required.

ELIGIBILITY:
Criteria:

* Histologically and/or cytologically confirmed malignant pleural mesothelioma.
* Unresectable disease (defined as the participant not being a candidate for curative surgery).
* Measurable disease, defined as at least 1 lesion (measurable) that can be accurately assessed at baseline by computed tomography (CT) or magnetic resonance imaging (MRI) and is suitable for repeated assessment (modified RECIST for pleural mesothelioma).
* Available unstained archived tumor tissue sample in sufficient quantity to allow for analyses. At least fifteen unstained slides or a tumor block (preferred). NOTE: A fine needle aspiration sample is not sufficient to make the patient eligible for enrollment. Given the complexity of mesothelioma pathological diagnosis and that these will be newly diagnosed patients it is expected that they will have a core needle biopsy or surgical tumor biopsy as part of their initial diagnostic work up.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Ability to understand and willingness to sign Institutional Review Board (IRB)-approved informed consent.
* Willing to provide archived tumor tissue and blood samples for research.
* Adequate organ function as measured by the following criteria, obtained ≤ 2 weeks prior to registration:

  * Absolute Neutrophil Count (ANC) ≥ 1500/mm³
  * Hemoglobin ˃9.0 g/dL
  * Platelets ˃100,000/mm³
  * Serum creatinine clearance (CL)>60 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance. NOTE: Patients with a creatinine Cl ≥ 45 mL/min however ≤ 60 mL/min may be considered for enrollment provided they fulfill all other eligibility criteria, these subjects will receive pemetrexed carboplatin concurrent with durvalumab during the combination phase of treatment. Patients with a creatinine CL<45 mL/min should not be enrolled.
  * Albumin ≥ 2.8 g/dL
  * Total Bilirubin ≤ 1.5x Upper Limit of Normal (ULN)
  * Aspartate Aminotransferase (AST)/Alanine Aminotransferase (ALT) ≤ 2.5x ULN (≤ 5x ULN in patients with liver metastases)
* Women must either be of non-reproductive potential or must have a negative serum pregnancy test upon study entry.
* Women must not be pregnant or breastfeeding.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up.
* Patient must not have involvement in the planning and/or conduct of the study. No previous enrollment in the present study.
* Patients may not have participated in another clinical study with an investigational product during the last 4 weeks.
* Patients must not have any prior systemic therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, and other investigational agent) for mesothelioma.
* No previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab or any other agent targeting immune checkpoints.
* Patients must not have non-pleural mesothelioma e.g. mesothelioma arising in peritoneum, tunica vaginalis or any serosal surface other than the pleura.
* Patients must not have an active second malignancy other than non-melanoma skin cancer or cervical carcinoma in situ.
* Patients must not have mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction.
* Patients must not have symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids (prednisone >10 mg or equivalent). Surgery, radiation and/or corticosteroids (any dose >10 mg prednisone equivalent) must have been completed ≥ 2 weeks prior to registration.
* Patients must not have uncontrolled seizures.
* Patients must not have current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Standard steroid premedication given prior to chemotherapy or as prophylaxis for imaging contrast allergy should not be counted for this criterion.
* No active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease, diverticulitis with the exception of diverticulosis, celiac disease, irritable bowel disease; Wegner syndrome) within the past 2 years. Subjects with vitiligo, alopecia, Grave's disease, or psoriasis not requiring systemic treatment (within the past 3 years) are not excluded.
* No history of primary immunodeficiency.
* No history of allogeneic organ transplant.
* No history of hypersensitivity to durvalumab, cisplatin, carboplatin, pemetrexed or any of their excipients.
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* No active infection including tuberculosis (clinical evaluation including: physical examination findings, radiographic findings, positive PPD test, etc.), hepatitis B (known positive HBV surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies as defined by a positive ELISA test). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. HIV testing is not required in absence of clinical suspicion.
* No known history of leptomeningeal carcinomatosis.
* Patients must not have received live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab.
* Patients must not have any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2020-02-16 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Forde, MD, Study Chair — John Hopkins
Locations (20):
- United States (20):
  - University San Diego Moores Cancer Center, La Jolla, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Stanford Cancer Institute, Stanford, California
  - University of Colorado, Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Miami Hospital, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Washington University in St Louis, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York University Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Hillman Cancer Center Research Pavilion, Pittsburgh, Pennsylvania
  - UTSW Medical Center, Dallas, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington
  - Aurora Cancer Center, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Data is proprietary.

REFERENCES:
- [Result] Forde PM, Anagnostou V, Sun Z, Dahlberg SE, Kindler HL, Niknafs N, Purcell T, Santana-Davila R, Dudek AZ, Borghaei H, Lanis M, Belcaid Z, Smith KN, Balan A, White JR, Cherry C, Ashok Sivakumar IK, Shao XM, Chan HY, Singh D, Thapa S, Illei PB, Pardoll DM, Karchin R, Velculescu VE, Brahmer JR, Ramalingam SS. Durvalumab with platinum-pemetrexed for unresectable pleural mesothelioma: survival, genomic and immunologic analyses from the phase 2 PrE0505 trial. Nat Med. 2021 Nov;27(11):1910-1920. doi: 10.1038/s41591-021-01541-0. Epub 2021 Nov 8. PMID 34750557
- [Derived] Kindler HL. Understanding the new therapeutic options for mesothelioma. Lancet Oncol. 2021 Oct;22(10):1353-1355. doi: 10.1016/S1470-2045(21)00520-9. Epub 2021 Sep 6. No abstract available. PMID 34499875

RESULTS

PARTICIPANT FLOW:
Groups:
- Concurrent Durvalumab Then Maintenance Durvalumab: Pemetrexed/cisplatin will be given for up to six 3-week cycles with the addition of concurrent durvalumab every 3 weeks. Use of carboplatin in place of cisplatin will be permitted for patients who are ineligible for cisplatin due to impaired renal function at screening. For patients that receive cisplatin, carboplatin may also be substituted after Cycle 1 for cisplatin related toxicity at the investigator's discretion.
  Concurrent Durvalumab: On Day 1 of each 21 day cycle: Durvalumab 1120 mg IV will be administered before pemetrexed and cisplatin chemotherapy over approximately 60 minutes. Approximately 30 minutes after the durvalumab infusion is complete, pemetrexed 500 mg/m² IV will be administered over 10 minutes. Cisplatin 75 mg/m² IV over 2 hours will begin approximately 30 minutes after the end of pemetrexed administration. If carboplatin is substituted for cisplatin, carboplatin Area Under the Concentration-Time Curve (AUC) 5 will be infused over 30 minutes beginning approximately 15-30 minutes after the end of the pemetrexed administration.
  After completion of Cycle 6 of concurrent therapy, patients with stable or responding disease per modified RECIST for malignant mesothelioma will continue on single agent durvalumab every 3 weeks until progression. Maximum duration of durvalumab treatment is 12 months starting from Cycle 1 of concurrent treatment.
  Maintenance Durvalumab: On Day 1 of each 21 day cycle: Durvalumab 1120 mg IV over approximately 60 minutes.
Period: Concurrent Durvalumab
Arm/Group | Concurrent Durvalumab Then Maintenance Durvalumab
Started | 55
Completed | 44
Not Completed | 11
Not completed — Adverse Event | 4
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Progressive Disease | 5
Period: Maintenance Durvalumab
Arm/Group | Concurrent Durvalumab Then Maintenance Durvalumab
Started | 44
Completed | 10
Not Completed | 34
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Progressive Disease | 31

BASELINE CHARACTERISTICS:
Arm/Group | Concurrent Durvalumab Then Maintenance Durvalumab
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 47
  More than one race | 0
  Unknown or Not Reported | 4
Histologic subtype [Count of Participants; unit: Participants]
  Epithelioid | 41
  Sarcomatoid | 7
  Biphasic | 6
  Desmoplastic | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from randomization to death from any cause. Patients that have not had an event reported at analysis will be censored at their date of last follow-up.
Time Frame: From randomization until death, up to 32 months
Population: All eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Concurrent Durvalumab Then Maintenance Durvalumab
Number analyzed (Participants) | 55
months | 20.4 [13.0 to 28.5]

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.03
Description: Number of participants with abnormal laboratory values and/or adverse events related to treatment.
Time Frame: Up to 15 months from start of treatment
Population: treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent Durvalumab Then Maintenance Durvalumab
Number analyzed (Participants) | 55
Participants | 36

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from randomization to documented disease progression or death from any cause, whichever occurs first. Patients who have not experienced an event of interest by the time of analysis will be censored at the date they are last known to be alive and progression-free.
Time Frame: From randomization until disease progression or death from any cause, up to 32 months
Population: Eligible and treated population
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Concurrent Durvalumab Then Maintenance Durvalumab
Number analyzed (Participants) | 55
month | 6.7 [6.1 to 8.4]

4. Secondary Outcome: Time to Progression (TTP) on Durvalumab
Description: TTP measured from the time concurrent treatment with chemotherapy/durvalumab begins until radiologic or clinical progression is noted.
Time Frame: From time concurrent treatment started until progression, up to 32 months
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Concurrent Durvalumab Then Maintenance Durvalumab
Number analyzed (Participants) | 55
months | 6.8 [6.2 to 8.4]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR assessed in accordance with RECIST 1.1 (modified for malignant mesothelioma).
Time Frame: From randomization until end of treatment, up to 15 months
Population: Eligible and treated patient population
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent Durvalumab Then Maintenance Durvalumab
Number analyzed (Participants) | 55
Participants | 31

ADVERSE EVENTS:
Time Frame: Adverse Events monitored for up to 15 months from start of treatment; deaths monitored from randomization for up to 32 months
Arm/Group | Concurrent Durvalumab Then Maintenance Durvalumab
All-Cause Mortality (participants affected / at risk) | 33/55
Serious Adverse Events (participants affected / at risk) | 36/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent Durvalumab Then Maintenance Durvalumab (N=55)
Anaemia (Blood and lymphatic system disorders) | 11 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Cellulitis (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Amylase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Confusional state (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Embolism (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (3)
Hypertensive emergency (Vascular disorders) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent Durvalumab Then Maintenance Durvalumab (N=55)
Anaemia (Blood and lymphatic system disorders) | 20
Hyperthyroidism (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 8
Dry eye (Eye disorders) | 7
Lacrimation increased (Eye disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 27
Diarrhoea (Gastrointestinal disorders) | 13
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 31
Vomiting (Gastrointestinal disorders) | 13
Asthenia (General disorders) | 3
Fatigue (General disorders) | 33
Mucosal inflammation (General disorders) | 3
Oedema peripheral (General disorders) | 9
Pyrexia (General disorders) | 7
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 6
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 3
Blood creatinine increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 3
Weight decreased (Investigations) | 9
Decreased appetite (Metabolism and nutrition disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 10
Hyponatraemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 8
Headache (Nervous system disorders) | 6
Memory impairment (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 5
Paraesthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 4
Confusional state (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 8
Acute kidney injury (Renal and urinary disorders) | 3
Dysuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 3
cough (Respiratory, thoracic and mediastinal disorders) | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Reproductive system and breast disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10
Upper-airway cough syndrome (Reproductive system and breast disorders) | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 11
Rash pruritic (Skin and subcutaneous tissue disorders) | 3
Hot flush (Vascular disorders) | 3
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT02899195/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT02899195/SAP_001.pdf